CLINICAL TRIAL: NCT03585751
Title: A Comparative Clinical and Radiographic Study of 3Mixstatin vs Tri-Antibiotic Mix and Simvastatin in the Treatment of Primary Molars With Inflammatory Root Resorption A Randomized Clinical Trial
Brief Title: 3Mixstatin ,Tri-Antibiotic Mix & Simvastatin in the Treatment of Primary Molars
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Dina El Kharadly, Assistant lecturer, October 6 University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3Mixstatin
Record Dates: First submitted 2018-06-08; First posted 2018-07-13 (Actual); Last update posted 2018-07-13 (Actual); Status verified 2018-06

CONDITIONS: Tooth, Deciduous
Keywords: non vital; deciduous; 3mixstatin; simvastatin; triple antibiotic mix; 3 mix
MeSH Terms: interventions — Pulpectomy; Simvastatin

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Every participant will grasp an opaque sealed envelop from a box after diagnosis of the case. Being opaque and sealed ensures allocation concealment. Envelopes have been assigned to RN who is not involved in neither the diagnosis nor the treatment phases of the cases.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Triple antibiotic paste (Active Comparator): Pulpectomy for primary molars, triple antibiotic mix is used as obturating material mixed with Macrogol and Polyethylene glycol & small amount of Zinc oxide powder to obtain workable , radio opaque mix
  Interventions: Procedure: Pulpectomy for primary molars + triple antibiotic mix
- 3mixstatin (Experimental): Pulpectomy for primary molars, 3 Mixstatin ( mix of simvastatin and triple antibiotic mix ) is used as obturating material mixed with Macrogol and Polyethylene glycol & small amount of Zinc oxide powder to obtain workable , radio opaque mix
  Interventions: Procedure: Pulpectomy for primary molars + 3mixstatin
- simvastatin (Experimental): Pulpectomy for primary molars, simvastatin is used as obturating material mixed with Macrogol and Polyethylene glycol & small amount of Zinc oxide powder to obtain workable , radio opaque mix
  Interventions: Procedure: Pulpectomy for primary molars + simvastatin

INTERVENTIONS:
Procedure: Pulpectomy for primary molars + triple antibiotic mix — complete extirpation of infected pulp from primary molars. Following instrumentation and copious irrigation ,the root canals are filled with one of .Following instrumentation and copious irrigation ,the root canals are filled with a triple antibiotic mix mixed with a Carrier ( MP) as an obturating material
  Arms: Triple antibiotic paste
Procedure: Pulpectomy for primary molars + 3mixstatin — complete extirpation of infected pulp from primary molars. Following instrumentation and copious irrigation ,the root canals are filled with one of .Following instrumentation and copious irrigation ,the root canals are filled with 3mixstatin (triple antibiotic mix + simvastatin) as an obturating material mixed with a Carrier ( MP) as an obturating material
  Arms: 3mixstatin
Procedure: Pulpectomy for primary molars + simvastatin — complete extirpation of infected pulp from primary molars. Following instrumentation and copious irrigation ,the root canals are filled with simvastatin as mixed with a Carrier ( MP) as an obturating material
  Arms: simvastatin

SUMMARY:
The aim of this study is to determine whether the success rate of pulp therapy undergone on primary molars with signs and symptoms of odontogenic infection that may render them indicated for extraction will improve with the use of the Simvastatin alone, the Tri-Antibiotic Mix alone or when in combination together 3Mixstatin as a component in the root filling material.

DETAILED DESCRIPTION:
A clinical situation will often present itself where primary teeth under radiographic examination show inter-radicular or periapical root resorption, perforation of coronal third of roots and/or loss of bone support as a result of infective or inflammatory conditions. Pathologic root resorption is the most common cause of premature tooth loss in primary dentition. The reason for that may be the high content of undifferentiated mesenchymal cells, which may give rise to odontoclastic cells in response to either the caries process or the pulp-capping materials, resulting in the exaggerated inflammatory response and consequently internal resorption in primary teeth. It would make sense to utilize the rich supply of undifferentiated mesenchymal cells towards regeneration of remaining dental tissues.

Antibiotic Mix as an intracanal medicament

In recent years, the Cariology Research Unit of Niigata University School of Dentistry has developed the concept of lesion sterilization and tissue repair (LSTR) therapy that employed a mixture of antibacterial drugs for disinfection. Repair of damaged tissues can be expected if lesions are disinfected. This procedure uses a mixture of three antibacterial drugs (3Mix MP) as a root canal medicament to eliminate the remaining bacteria in endodontic lesions. The medicament consists of metronidazole, ciprofloxacin and minocycline - with macrogol (M) as the ointment base and propylene glycol (P) as the carrier Alone, none of these drugs resulted in complete elimination of the bacteria. However, in combination, these drugs were able to consistently sterilize all samples.

Although a local antibiotic medication in endodontics offers many advantages, this mode has some drawbacks, including development of bacterial resistant strains. That is a major concern and may lead to the transfer of resistance genes from antibiotic-resistant to antibiotic-susceptible microorganisms. Other drawbacks include allergic reactions inhibition of angiogenesis , and tooth staining or discoloration particularly with Minocycline. More importantly is that although the concept of Lesion sterilization and tissue repair (LSTR) therapy is that it provides an efficient and predictable disinfection, through 3 Mix on a local level and providing the suitable environment for tissues to heal, it does not in itself have any anti-inflammatory nor regenerative potential. Statins may provide these two benefit.

Choice of comparator Statins are structural analogs of HMG-CoA (3hydroxy-3-methylglutaryl-coenzyme A). These drugs are the first-line for hyperlipidemia and it has been recognized to be a safe and low-priced drug as a result of its worldwide longtime usage. Moreover, statins have multiple functions including anti-inflammation, induction of angiogenesis and improvement of the vascular endothelial cell function. Another interesting and important function of statin is its effect on bone formation. It has been reported that several statins such as simvastatin and lovastatin have anabolic effects on bone metabolism at in vitro and in vivo studies. They promote mineralization in non-mineralizing osteoblasts through induction of BMP-2 and osteocalcin. Local application of simvastatin gel has shown to stimulate the regeneration of alveolar bone defects Statins have an anti-inflammatory effect. They act by decreasing the production of interleukin-6 and interleukin-8 and may also improve the function of odontoblasts, thus dentin formation.

3 Mixstatin as an intracanal medicament

Often, different chemicals or drugs are combination in a cocktail in an attempt to elicit variety of effects with a single application.

Aminabadi et al combined the above-mentioned techniques by adding simvastatin powder to the tri-antibiotic mix (3Mix) and proposed the term "3Mixtatin", (an acronym of 3Mix and simvastatin) with the aims of suppressing bacteria, preventing pulp inflammation, and inducing hard tissue formation. His study population involved poor prognosis primary molars with advanced root resorption and/or pulpal floor perforation.

When compared with MTA, radio graphic and clinical healing occurred more successfully following 3Mixtatin treatment within a 24-month study period 96.8% success rate both clinically and radiographically. 3Mixstatin, a previously unstudied combination was applied, lead to preservation of the primary teeth that were otherwise indicated for extraction according to current guidelines. It may lead to a paradigm shift in the treatment of primary teeth in the future.

ELIGIBILITY:
Inclusion Criteria:

Patients:

1. Young cooperative patients with no history of systemic disease that may contraindicate pulp therapy
2. Age range 4-6 years.
3. Patient has at least one restorable primary molar that exhibits signs and symptoms of odontogenic infection with inflammatory root resorption and require pulpectomy,
4. Patient's parents are willing to participate in this study and will be able to follow up Clinical & Radiographic Criteria for Case Selection Signs and symptoms of irreversible pulpitis as well as inter-radicular, or periapical root resorption as a result of infective or inflammatory conditions that may render the tooth hopeless and indicated for extraction

Clinical Criteria (include):

1. Spontaneous pain
2. Intraoral Abscess
3. Extra oral Abscess
4. Tender to percussion
5. Presence of abnormal mobility other than that associated with exfoliation

Radiographic Criteria include:

1. Radiolucency in furcation area 2. Periapical root resorption or excessive bone destruction and/or perforation in coronal third of roots as a result of infective or inflammatory conditions.

-

Exclusion Criteria:

* Patients with systemic disease 2. Patients who cannot attend follow up. 3. Primary molars that are unrestorable 4. Primary molars exhibiting pathology of permanent tooth follicle

Ages: 5 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 45 (Estimated)
Dates: Start 2018-09 (Estimated); Primary Completion 2019-09 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Over All Success Rate ( as a percentage) | 12 months
  For each group
  Number of cases exhibiting success criterion at 12 months / Total number of cases x 100
  At the end of the follow up period, the cases are considered successful if they exhibited ALL the following criteria:
  * Absence of tenderness to percussion
  * No abnormal mobility
  * Absence of swelling and fistula
  * Absence or decrease of furcation radiolucency
  * Absence or decrease of radicular radiolucency
  * Absence of Internal/external root resorption or other pathological changes
  The cases were considered as total (overall) failures if they failed clinically at the 3, 6 or 12 months; or when they failed radiographically at the 12 months follow-up.
  Otherwise they will be considered as a success.

SECONDARY OUTCOMES:
Bone density changes in Region of Interest ROI | 12 months
  measured by :Digora image analysis software i.e. Digora for windows software DFW Measuring Unit :Relative pixel values using an 8-bit scale from full black (0) to full white (255)

CONTACTS AND LOCATIONS:
Overall Officials: Sherif B El Tawil, DDS, Study Chair — Cairo University; Dina El Beshlawy, Study Director — Cairo University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aminabadi NA, Huang B, Samiei M, Agheli S, Jamali Z, Shirazi S. A Randomized Trial Using 3Mixtatin Compared to MTA in Primary Molars with Inflammatory Root Resorption: A Novel Endodontic Biomaterial. J Clin Pediatr Dent. 2016;40(2):95-102. doi: 10.17796/1053-4628-40.2.95. PMID 26950808
- [Background] Takushige T, Cruz EV, Asgor Moral A, Hoshino E. Endodontic treatment of primary teeth using a combination of antibacterial drugs. Int Endod J. 2004 Feb;37(2):132-8. doi: 10.1111/j.0143-2885.2004.00771.x. PMID 14871180
- [Background] Asl Aminabadi N, Maljaei E, Erfanparast L, Ala Aghbali A, Hamishehkar H, Najafpour E. Simvastatin versus Calcium Hydroxide Direct Pulp Capping of Human Primary Molars: A Randomized Clinical Trial. J Dent Res Dent Clin Dent Prospects. 2013 Winter;7(1):8-14. doi: 10.5681/joddd.2013.002. Epub 2013 Feb 21. PMID 23487477
- [Background] Doneria D, Thakur S, Singhal P, Chauhan D, Keshav K, Uppal A. In Search of a Novel Substitute: Clinical and Radiological Success of Lesion Sterilization and Tissue Repair with Modified 3Mix-MP Antibiotic Paste and Conventional Pulpectomy for Primary Molars with Pulp Involvement with 18 Months Follow-up. Contemp Clin Dent. 2017 Oct-Dec;8(4):514-521. doi: 10.4103/ccd.ccd_47_17. PMID 29326499
- [Background] Nakornchai S, Banditsing P, Visetratana N. Clinical evaluation of 3Mix and Vitapex as treatment options for pulpally involved primary molars. Int J Paediatr Dent. 2010 May;20(3):214-21. doi: 10.1111/j.1365-263X.2010.01044.x. PMID 20409203
- [Background] Okamoto Y, Sonoyama W, Ono M, Akiyama K, Fujisawa T, Oshima M, Tsuchimoto Y, Matsuka Y, Yasuda T, Shi S, Kuboki T. Simvastatin induces the odontogenic differentiation of human dental pulp stem cells in vitro and in vivo. J Endod. 2009 Mar;35(3):367-72. doi: 10.1016/j.joen.2008.11.024. PMID 19249597
- [Background] Seto H, Ohba H, Tokunaga K, Hama H, Horibe M, Nagata T. Topical administration of simvastatin recovers alveolar bone loss in rats. J Periodontal Res. 2008 Jun;43(3):261-7. doi: 10.1111/j.1600-0765.2007.01024.x. PMID 18447852
- [Background] Chen S, Yang JY, Zhang SY, Feng L, Ren J. Effects of simvastatin gel on bone regeneration in alveolar defects in miniature pigs. Chin Med J (Engl). 2011 Dec;124(23):3953-8. PMID 22340324
- [Background] Sakoda K, Yamamoto M, Negishi Y, Liao JK, Node K, Izumi Y. Simvastatin decreases IL-6 and IL-8 production in epithelial cells. J Dent Res. 2006 Jun;85(6):520-3. doi: 10.1177/154405910608500608. PMID 16723648